CLINICAL TRIAL: NCT05700552
Title: The Effect of Skin-to-Skin Contact After Elective Cesarean Section on Pain and Stress Levels of the First Intramuscular Injection of the Newborn
Brief Title: Skin-to-skin Contact for Newborn First Injection Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Kocaeli University (Other)
Responsible Party: Principal Investigator, sena dilek, Principal Investigator, Kocaeli University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: sdilek3
Record Dates: First submitted 2023-01-06; First posted 2023-01-26 (Actual); Last update posted 2023-12-14 (Actual); Status verified 2023-12

CONDITIONS: Pain
Keywords: skin to skin contact; Newborn; stress; cesarean section
MeSH Terms: conditions — Pain | interventions — Kangaroo-Mother Care Method

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): In the intervention group, after cesarean delivery in the operating room, maternal vital signs and the newborn's 1st and 5th minute Apgar Score will be evaluated. After the newborn baby is aspirated if necessary, dried with a green cover under the radiant warmer, tied the diaper, and put on a hat, the newborn with an Apgar Score ≥7 and vital signs stable will be wrapped in pre-warmed operating room covers. After providing a suitable environment, the newborn whose body temperature is stabilized will be placed in the prone position without any covering and clothing on the chest area of the mother, and the ALPS value will be applied for about 3 minutes due to the application of hospital procedures, the intramuscular injection will be applied and the ALPS score will be evaluated again after the injection.
  Interventions: Behavioral: skin to skin contact
- Control group (No Intervention): The routine procedure of the institution where the study will be performed will be applied to the newborn baby after cesarean section in the control group. Within the scope of this procedure, after the baby is born, the umbilical cord is cut, mouth and nose aspiration is performed under the radiant heater in the operating room, they are dried, and the Apgar Score is evaluated at the 1st and 5th minutes by the midwife. The newborn is wrapped in pre-heated operating room covers, and after being shown to the mother, anthropometric measurements (height, body weight, head circumference) are taken and taken to the delivery room for the administration of vitamin K, hepatitis B vaccine, and the first examination of the baby. The first ALPS value will be recorded in the delivery room in the baby care area, the intramuscular injection will be applied and the ALPS score will be evaluated again after the injection.

INTERVENTIONS:
Behavioral: skin to skin contact — For skin-to-skin contact (TTT), the newborn is placed naked on the mother's bare chest in the prone (prone) position, the newborn's abdomen and chest are in contact with the mother's skin, and the newborn's head is turned to the side so that the airway remains open.
  Other Names: kangaroo care
  Arms: Intervention Group

SUMMARY:
This study is carried out to examine the effect of skin-to-skin contact on the pain and stress level of the first intramuscular injection after elective cesarean section. The universe of the research will be women who have had elective cesarean section at Darıca Farabi Training and Research Hospital. The sample size of the study was calculated using the G*Power 3.1.9.2 program. The minimum number of individuals to be included in the sample of this study was calculated by taking G*Power 3.1.9.2, effect size: 1.42 α= 0.05, power: 0.95, and the sample size was determined as at least 14 mothers and their newborns in each group (skin skin-to-skin contact group: 14, non-skin-to-skin contact group: 14). In the study, possible data losses will be foreseen and 60 newborns and mothers, 30 of which will be in the intervention group and 30 in the control group, will be taken. The group of the participants included in the research will be divided into two groups by determining the random number generation program on the website called "Random List". (https://www.randomlists.com/). After obtaining the necessary ethics committee and institutional permissions for the implementation of the study, participants who had a cesarean delivery and who met the inclusion criteria of the study will be interviewed by going to the institution. Those who accept and want to participate in the research will have the Voluntary Consent Form read and their signatures will be taken. Term newborns meeting the criteria will be divided into intervention and control groups. The data will be collected by the researcher working in the delivery room of the hospital through face-to-face interviews. In the study, newborns who received skin-to-skin contact during the first IM injection will be included in the intervention group, and newborns who have been routinely injected intramuscularly in the delivery room will be included in the control group. In the study, all the steps of the intervention and control group newborns before and after the application will be carried out by the researcher.

DETAILED DESCRIPTION:
Aim: This study will be carried out to examine the effect of skin-to-skin contact after elective cesarean section on the pain and stress level of the first intramuscular injection given to the newborn.

Research hypothesis:

Hypothesis (H0): Skin-to-skin contact has no effect on the level of pain and stress felt during the first intramuscular injection in newborns after elective cesarean section.

Hypothesis (H1): Skin-to-skin contact has an effect on the level of pain and stress felt during the first intramuscular injection in newborns after elective cesarean section.

Type of Study: This study was designed as a randomized controlled experimental study.

Data will be collected by the researcher from the Delivery Room and Operating Room units. Before the skin-to-skin contact procedure after elective cesarean section, the mother will be informed about the application and the purpose of the research will be explained. Those who accept and want to participate in the research will have the Voluntary Consent Form read and their signatures will be taken. Term newborns meeting the criteria will be divided into intervention and control groups. In determining the selection process, the random number generation program will be divided into two groups by using the website called "Random List". (https://www.randomlists.com/). Thus, each participant's group and group number will be determined and recorded. In the study, newborns who received skin-to-skin contact during the first IM injection will be included in the intervention group, and newborns who have been routinely injected intramuscularly in the delivery room will be included in the control group. In the study, all the steps of the intervention and control group newborns before and after the application will be carried out by the researcher.

Research data will be collected by using the Pregnancy Information Form, Neonatal Follow-up Form and Neonatal Pain and Stress Assessment Scale (ALPS-Neo) created by the researchers within the framework of the relevant literature.

Pregnant Information Form: It was prepared by the researcher within the framework of the literature. The form consists of a total of 19 questions, 7 open-ended and 12 closed-ended, questioning women's socio-demographic knowledge of obstetrics.

Neonatal Follow-up Form: Newborn's vital sign measurements (body temperature, blood pressure, heart rate, oxygen saturation, respiratory rate), orocephalic response (head orientation, sucking reflex, oral movement, facial expression) and first breastfeeding initiation, including newborn introductory features. It contains 26 questions consisting of a table in which time and duration measurements will be recorded.

Neonatal pain and stress rating scale (ALPS-Neo): Lundqvist et al. (2014) to evaluate pain and stress in premature and term newborns. The Cronbach's alpha coefficient of the scale was reported as 0.95. The scale is a 0-1-2, 3-point Likert type scale consisting of 5 items in one dimension, including the newborn's facial expression, breathing pattern, tone of the extremities, hand and foot activities, and activity level. Measurements are made by observation. A minimum of 0 and a maximum of 10 points are obtained from the scale. As a result of the evaluation, 3-5 points indicate the presence of mild pain and stress, and more than 5 points indicate the presence of severe pain and stress. The higher the stress and pain, the higher the score.

Applicable to the Intervention Group In the intervention group, after cesarean delivery in the operating room, maternal vital signs and the newborn's 1st and 5th minute Apgar Score will be evaluated. After the newborn baby is aspirated if necessary, dried with a green cover under the radiant warmer, tied the diaper, and put on a hat, the newborn with an Apgar Score ≥7 and vital signs stable will be wrapped in pre-warmed operating room covers. Preheated blankets will be placed on the chest area of the mother in the same way and her temperature will be measured with a thermometer before skin-to-skin contact. Those with low body temperature will be excluded. After providing a suitable environment, the newborn whose body temperature is stabilized will be placed in the prone position without any covering and clothing on the chest area of the mother, and due to the implementation of hospital procedures, skin-to-skin contact will be applied for about 3 minutes and the first injection will be performed. After the injection, vital signs of the newborn (body temperature, blood pressure, peak heart rate, oxygen saturation, respiratory rate) will be measured, oxygen demand, orocephalic responses (head orientation, sucking reflex, oral movement, facial expression) will be observed, ALPS-Neo Newborn Pain and the scores from the Stress Rating Scale will be evaluated and recorded. Further examinations of the newborn will take place in the delivery room. When the mother is transferred from the operating room to the gynecology service, her newborn will be taken. And the time and duration of first breastfeeding initiation will be evaluated and recorded.

Applicable to the Control Group The routine procedure of the institution where the study will be performed will be applied to the newborn baby after cesarean section in the control group. Within the scope of this procedure, after the baby is born, the umbilical cord is cut, mouth and nose aspiration is performed under the radiant heater in the operating room, they are dried, and the Apgar Score is evaluated at the 1st and 5th minutes by the midwife. The newborn is wrapped in pre-heated operating room covers, and after being shown to the mother, anthropometric measurements (height, body weight, head circumference) are taken and taken to the delivery room for the administration of vitamin K, hepatitis B vaccine, and the first examination of the baby. After the injection, vital signs of the newborn (body temperature, blood pressure, peak heart rate, oxygen saturation, respiratory rate) will be measured, oxygen demand, orocephalic responses (head orientation, sucking reflex, oral movement, facial expression) will be observed, ALPS-Neo Newborn Pain and the scores from the Stress Rating Scale will be evaluated and recorded. After the newborn's procedures and examination, he is transferred to his room in the gynecology service. On average, these processes and transfer time take 30-45 minutes. As a routine practice of the hospital, due to the transfer process and stabilization of the patient, the first skin contact of the mother and the baby and the time to start breastfeeding take place approximately 1-2 hours later. This process will be observed and the first breastfeeding time will be recorded by evaluating the skin-to-skin contact time and breastfeeding time.

Statistical and Analytical Methods:

Statistical analysis will be performed using the IBM SPSS Statistic 22.0 (IBM Corp. , Armonk , NY, USA) program. Descriptive statistical methods (number, percentage, mean, standard deviation) will be used in the evaluation of sociodemographic data. Parametric tests (chi-square, T test, etc.) and non-paramedic tests (Mann-Whitney U Test, Kruskal Wallis, etc.) will be used in the comparison of categorical variables when it is seen that the data are suitable for normal distribution) will be used when it is not suitable for a normal distribution. P significance level will be accepted as 0.05.

ELIGIBILITY:
Inclusion Criteria:

* Able to speak and understand Turkish,
* Conceiving naturally,
* At the end of the gestational week (37-42 weeks),
* Will have an elective cesarean delivery,
* In cesarean delivery, only spinal anesthesia is applied,
* No hearing problem,
* Women willing to participate in the research,
* Not having a risky pregnancy,
* Single fetus,
* A first-minute APGAR score (scoring system that shows the newborn's health status) is 7 and above (healthy newborn that does not require any intervention),
* No congenital anomaly,
* Does not require observation in neonatal intensive care,
* Newborns with a birth weight between 2500 - 4000 g.

Exclusion Criteria:

* Those who do not have sufficient mental health to fill out the questionnaire,
* Newborns who need oxygen support or dead newborns
* Exposed to any painful stimulus (Venous-capillary sample),
* Those who may refuse to receive the hepatitis B vaccine, vitamin K or any injections
* Women and newborns with any maternal and/or neonatal risk conditions in the early postpartum period will not be included in the study.

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes
Enrollment: 60 (Actual)
Dates: Start 2023-01-06 (Actual); Primary Completion 2023-05-31 (Actual); Study Completion 2023-07-18 (Actual)

PRIMARY OUTCOMES:
ALPS-Neo Neonatal Pain and Stress Rating Scale | This scala will be evaluated just before the intramuscular injection.
  The scale is a 0-1-2, 3-point Likert type scale consisting of 5 items in one dimension, including the newborn's facial expression, breathing pattern, tone of the extremities, hand and foot activities, and activity level. Measurements are made by observation. A minimum of 0 and a maximum of 10 points are obtained from the scale. As a result of the evaluation, 3-5 points indicate the presence of mild pain and stress, and more than 5 points indicate the presence of severe pain and stress. The higher the stress and pain, the higher the score.
ALPS-Neo Neonatal Pain and Stress Rating Scale | This scala will be evaluated after administering the intramuscular injection.
  The scale is a 0-1-2, 3-point Likert type scale consisting of 5 items in one dimension, including the newborn's facial expression, breathing pattern, tone of the extremities, hand and foot activities, and activity level. Measurements are made by observation. A minimum of 0 and a maximum of 10 points are obtained from the scale. As a result of the evaluation, 3-5 points indicate the presence of mild pain and stress, and more than 5 points indicate the presence of severe pain and stress. The higher the stress and pain, the higher the score.

CONTACTS AND LOCATIONS:
Overall Officials: Sena Dilek Aksoy, Ph.D, Study Director — Kocaeli University; Seda Yazici, M.Sc., Study Chair — Kocaeli Darica Farabi Training and Research Hospital
Locations (1):
- Kocaeli University, Kocaeli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No